CLINICAL TRIAL: NCT06783387
Title: Physical Activity, Mediterranean Diet and Maternity Blues: a Multidisciplinary Approach
Acronym: MMB/01
Status: Not yet recruiting | Type: Observational
Sponsor: Centro Universitario Ricerca Interdipartimentale Attivita' Motoria (Other)
Collaborators: Sezione di Psichiatria Psicologia Clinica e Riabilitazione del Dipartimento di Medicina e Chirurgia dell'Università degli Studi di Perugia (Unknown); Scuola di Specializzazione in Ginecologia ed Ostetricia del Dipartimento di Medicina e Chirurgia dell' Università degli Studi di Perugia. (Unknown); Sezione di Clinica Ostetrica e Ginecologia del Dipartimento di Medicina e Chirurgia dell' Università degli Studi di Perugia (Unknown); Clinica Ostetrica Ginecologica dell'Università degli Studi di Palermo (Unknown); Scuola di Specializzazione in Psichiatria del Dipartimento di Medicina dell'Università degli Studi di Perugia (Unknown); Centro Universitario Ricerca Interdipartimentale Attivita' Motoria del Dipartimento di Medicina dell''Università degli Studi di Perugia (Unknown)
Responsible Party: Sponsor
Other Study IDs: CURicerca
Record Dates: First submitted 2024-12-12; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Maternity Blues
Keywords: maternity blues; Physical activity; multidisciplinary approach; Mediterranean diet
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- New mothers: 544 women who have recently given birth in one of the Clinics involved in the study will be invited to respond to an online questionnaire.

SUMMARY:
This study aims to evaluate the levels of physical activity, sedentary time, eating habits, and emotional well-being in a group of women after giving birth.

DETAILED DESCRIPTION:
The study involves the enrollment of 544 subjects and the overall expected duration is 24 months.

The study is observational, as it only involves collecting and recording information and clinical data according to the times and methods of treatment to which women are subjected in normal hospital practice.

In particular, the collection of information about:

* general nature;
* the pregnancy;
* participants' levels of physical activity and sedentary lifestyle;
* participants' nutritional habits;
* factors that influence participants' emotional well-being. The data will be collected in digital format, through filling out an online questionnaire. The data obtained will be organized in a digital file and processed in aggregate and anonymous form. Access to the data will be permitted only to personnel authorized for the study.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects, aged ≥18 years and with adequate knowledge of spoken and written Italian.

Exclusion Criteria:

* Presence of pathologies that contraindicate the practice of physical activity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Puerperal women within three days of giving birth who decide to participate, voluntarily, autonomously and anonymously, in the survey via an online questionnaire, according to non-probability convenience sampling.
Sampling Method: Non-Probability Sample
Enrollment: 544 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Levels and sedentary time | From the moment of enlistment and within the first 10 days after giving birth
  Physical Activity Levels and sedentary time data will be collected using the l'International Physical Activity Questionnaire
Mediterranean Diet Adherence | From the moment of enlistment and within the first 10 days after giving birth
  Mediterranean Diet Adherence data will be collected using the 14-item Mediterranean diet assessment tool
Presence of symptoms of maternity blues | From the moment of enlistment and within the first 10 days after giving birth
  These data will be collected using the Edinburgh Postnatal Depression Scale
Date of birth | The questionnaire will be proposed within the first 10 days after giving birth
  Number of days since giving birth

SECONDARY OUTCOMES:
City of birth | At the moment of enlistment
  indicate in which city you gave birth
Degree | From the moment of enlistment
  Degree (choose from):
  * Primary school
  * Middle school (or lower secondary school)
  * Secondary school (or upper secondary school)
  * Bachelor's degree
  * PhD/Specialization
Marital status | At the moment of enlistment
  Marital status, choosing from:
  * Single.
  * Cohabiting/Married.
  * Separated/Divorced.
  * Widow.
Age | At the moment of enlistment
  Age, in years
Weight before pregnancy | before pregnancy
  Weight in kilograms
Weight at the moment of enlistment | At the moment of enlistment
  Weight in kilograms
height | At the moment of enlistment
  height in meters

OTHER OUTCOMES:
Information about pregnancy and state of health | At the moment of enlistment
  Some closed questions were proposed to ask the participants if they had other pregnancies before this one (operative births, spontaneous births, spontaneous abortions, etc...); if they had previously suffered from Postpartum Depression Maternity blues Postpartum psychosis, and if during this pregnancy one or more pathologies were diagnosed (for example Gestational Diabetes, Gestational Hypertension, etc...)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Favilli, Principal Investigator — Sezione di Clinica Ostetrica e Ginecologia del Dipartimento di Medicina e Chirurgia dell' Università degli Studi di Perugia; Giulia Menculini, Principal Investigator — Sezione di Psichiatria Psicologia Clinica e Riabilitazione del Dipartimento di Medicina e Chirurgia dell'Università degli Studi di Perugia; Roberto Pippi, Principal Investigator — Centro Universitario Ricerca Interdipartimentale Attivita' Motoria del Dipartimento di Medicina e Chirurgia dell' Università degli Studi di Perugia
Locations (5):
- Italy (5):
  - Centro Universitario Ricerca Interdipartimentale Attivita' Motoria del Dipartimento di Medicina dell''Università degli Studi di Perugia, Perugia, Italy
  - Clinica Ostetrica e Ginecologica dell' Azienda Ospedaliera di Perugia, Perugia, Italy
  - Scuola di Specializzazione in Ginecologia ed Ostetricia del Dipartimento di Medicina e Chirurgia dell' Università degli Studi di Perugia, Perugia, Italy
  - Scuola di Specializzazione in Psichiatria del Dipartimento di Medicina dell'Università degli Studi di Perugia, Perugia, Italy
  - Sezione di Psichiatria, Psicologia Clinica e Riabilitazione Psichiatrica del Dipartimento di Medicina e Chirurgia dell' Università degli Studi di Perugia., Perugia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF